CLINICAL TRIAL: NCT06195020
Title: Examining the Effect of Metaverse-Based Epilepsy Education on Parents' Epilepsy Knowledge Level: Randomized Controlled Experimental Research
Brief Title: Examining the Effect of Metaverse-Based Epilepsy Education
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Mehmet Duray, Assist Prof, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 72867572-050.01.04
Record Dates: First submitted 2023-12-21; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Examining the Effect of Metaverse-based Epilepsy Education on Parents' Knowledge Level
Keywords: Epilepsy; metaverse; parent; knowledge level
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): This group will be informed by sharing and using educational videos prepared in the Metaverse universe on mobile.
  Interventions: Other: Metaverse
- Control Group (Active Comparator): This group will be informed through routine outpatient clinic service.
  Interventions: Other: Polyclinic information

INTERVENTIONS:
Other: Metaverse — The research consists of two stages (preparation and implementation). In the first stage of the research, the educational material planned to be used in the education of parents (video of navigation in the metaverse) will be developed in the form of modules. The topics in the training materials to be developed are listed below.
  Module 1: Information about Epilepsy (What is epilepsy?, What are the causes of epilepsy? Module 2 Diagnostic Methods in Epilepsy (Neurological examination, blood tests, electroencephalogram, screening tests 3rd Module Treatment of Epilepsy (Things to consider in patients receiving antiepileptic drug therapy) Module 4: First Aid in Epilepsy (first aid in seizures with convulsions, first aid in seizures without convulsions) Module 5: Life with Epilepsy (Epilepsy and school, epilepsy and career choice, epilepsy and home safety, epilepsy and exercise, epilepsy and healthy nutrition, epilepsy and sleep) The intervention will last 3 months.
  Arms: Experimental Group
Other: Polyclinic information — This group will be informed only at the outpatient clinic. The intervention will last 3 months.
  Arms: Control Group

SUMMARY:
The research is a randomized controlled experimental study and was planned to examine the effect of metaverse-based epilepsy education on the epilepsy knowledge level of parents.

DETAILED DESCRIPTION:
Developments in the field of technology, patient density in polyclinic services, limited number of nurses specialized in the field and the desire to carry out effective workforce planning bring different education methods to the agenda in the field of nursing. Creating the metaverse universe, which has been used in many technological fields in recent years, is among the newest of these technological developments. When the content created in Metaverse-based training is presented to the user, the user has the opportunity to enter the universe, choose the avatar the participant wants, and navigate and gain information by entering the desired module among the training modules created for participant. At the same time, since it offers an interactive training module to the participant, there are no limitations such as time, place or subject as in other training models. When the literature was examined, no study was found in which metaverse-based education was used in the field of epilepsy. In this context, our research aimed to examine the usability of metaverse-based epilepsy education and its effect on parents' epilepsy knowledge level.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to use a smartphone with internet access
* Having a child diagnosed with epilepsy

Exclusion Criteria:

* Having an additional chronic disease (diabetes, chronic kidney failure, cancer, etc.) other than epilepsy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Introductory Form Regarding Parents and the Child's Illness | 3 months
  This form consists of 9 questions and includes descriptive characteristics of the parents (age, mother/father, education level) and information about the epilepsy disease (mother/father age, educational status, occupation, diagnosis). questions (time, medications used, sources of information about the disease).
Epilepsy Knowledge Test Developed for Parents | 3 months
  This test, developed by researchers in line with the literature, consists of 50 questions. Answers to each test question can be given as "true", "false" or "I don't know".

SECONDARY OUTCOMES:
Application Content and Quality Evaluation by the Expert Group [DISCERN Measurement Tool (Quality of Criteria for Consumer Health Information)] | 3 months
  The DISCERN measurement tool was developed by Charnock et al. (1999) to be used in evaluating the content and quality of the educational material. The DISCERN measurement tool, which consists of three parts, contains 16 questions that question the content of the material. The first part, consisting of eight questions, measures the reliability of the material, the second part, consisting of seven questions, measures the quality of the information provided on treatment/care options, while the third part, consisting of a single question, questions the general evaluation of the material. In DISCERN, each question is scored from 1 to 5, where "5" indicates the suitability of the material and "1" indicates the inappropriateness of the material. By summing the responses from each item, a score between 15 and 75 is obtained. Article 16, which gives the general evaluation, is evaluated separately.
System Usability Scale (SUS) | 3 months
  This measurement tool will be applied to parents in evaluating the usability of the developed universe. Created by John Brooke in 1986, this scale allows evaluation of a wide range of products and services, including hardware, software, mobile devices, websites and applications. Five-point Likert-type scale consisting of 10 items. The scale consists of 10 items and has a 5-point Likert-type evaluation (0: strongly disagree, 1: disagree, 2: undecided, 3: agree, 4: strongly agree). Items 2, 4, 6, 8 and 10 in the scale are scored in reverse, and the score obtained from each participant is multiplied by 2.5 to obtain a score between 0-100. Based on research, an SUS score above 68 is considered above average and any score below 68 is considered below average (https://www.usability.gov/how-to-and-tools/methods/system-usability -scale.html Access Date: 28.02.2021).

CONTACTS AND LOCATIONS:
Locations (1):
- Mehmet Duray, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No